CLINICAL TRIAL: NCT01315821
Title: Role Of Saccharomyces Boulardii in Preventin Necrotizing Enterocolitis in Very Low Birth Weight Infants
Brief Title: Effect of Saccharomyces Boulardii on Necrotizing Enterocolitis in Very Low Birth Weight Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity Teaching Hospital, Zekai Tahir Burak Maternity Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1234
Record Dates: First submitted 2011-02-24; First posted 2011-03-15 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-02

CONDITIONS: Necrotizing Enterocolitis; Very Low Birth Weight Infants
Keywords: Saccharomyces boulardii; necrotizing enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saccharomyces boulardii (Experimental): Saccharomyces boulardii 5 million unit/day for 3 months
  Interventions: Drug: Saccharomyces boulardii
- control (Placebo Comparator): Placebo- for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saccharomyces boulardii — 5 million units/day for 3 months
  Other Names: Reflor
  Arms: Saccharomyces boulardii
Drug: Placebo — Placebo for 3 months
  Arms: control

SUMMARY:
Probiotics are favorable microorganisms that regulate the flora of the gastrointestinal system and stimulate the immune system. Necrotizing enterocolitis incidence is 10-25% in newborn infants whose birth weights are < 1500 gr. Although bifidobacterium and lactobacilli sp. have been used to reduce the incidence of NEC in clinical trials, Saccharomyces boulardii has not been used in the prevention of NEC in very low birth weight infants yet. The objective of this study is to evaluate the efficacy of orally administered S boulardii in reducing the incidence and severity of NEC in very low birth weight infants.

DETAILED DESCRIPTION:
The primary outcome of this study is to evaluate the efficacy of orally administered S boulardii in reducing the incidence and severity of NEC in very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants < 1500 gr

Exclusion Criteria:

* Genetic anomalies
* Not willing to participate
* Allergy to S. boulardii components

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Effect of Saccharomyces boulardii on necrotizing enterocolitis in VLBW infants | up to 6 months

SECONDARY OUTCOMES:
Effect of Saccharomyces boulardii on culture proved sepsis | 6 months
Effect of Saccharomyces boulardii on weight gain | up to 6 months
Effect of Saccharomyces boulardii on length of hospital stay | up to 6 months
Effect of Saccharomyces boulardii on mortality | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Demirel, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD005496. doi: 10.1002/14651858.CD005496.pub6. PMID 37493095
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD005496. doi: 10.1002/14651858.CD005496.pub5. PMID 33058137